CLINICAL TRIAL: NCT03076242
Title: Genetic Evaluation of Men (GEM)
Status: Terminated | Type: Observational
Why Stopped: Competing trial
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Myriad Genetics, Inc. (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Other Study IDs: 14S.546; JT 6981 (Other: JeffTrial Number)
Record Dates: First submitted 2017-03-06; First posted 2017-03-10 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gem Registry: Men with a personal history of PCA; Unaffected males who are at higher risk for prostate cancer
  Interventions: Other: GEM Registry

INTERVENTIONS:
Other: GEM Registry — Men with a personal history of PCA; Unaffected males who are at higher risk for prostate cancer

SUMMARY:
This is a prospective research registry and prospective genetic testing cohort study. The goal is to collect personal medical and cancer history data, family cancer data, exposure history, and biospecimens to support research focused on optimal genetic testing strategies for men with prostate cancer with the ultimate goal of informing national guidelines focused on genetic evaluation for prostate cancer.

DETAILED DESCRIPTION:
Objectives:

1. Collect detailed family cancer histories, personal medical history, prostate cancer clinical features, and exposure history from men with prostate cancer and men without prostate cancer to support studies focused on identifying hereditary cancer syndromes and genetic/epidemiologic factors predisposing to prostate cancer susceptibility.
2. Collect behavioral measures to support research focused on assessing the needs of men undergoing cancer risk evaluation and satisfaction with the process.
3. Create and maintain a biospecimen bank with specimens from men with prostate cancer and without prostate cancer to support studies focused on genetic alterations predisposing to prostate cancer risk.
4. Perform targeted and broad-scale genetic and genomic sequencing to detect genetic alterations related to prostate cancer risk.
5. Develop mechanisms to recontact participants with updates on research genetic results to guide genetic testing for inherited prostate cancer risk.

ELIGIBILITY:
Inclusion Criteria:

1. Men with a personal history of prostate cancer
2. Unaffected males who are at higher risk for prostate cancer

Exclusion Criteria:

1. Age < 18 years
2. Mental or cognitive impairment that interferes with ability to provide informed consent
3. Social circumstances that may impair the ability to follow through with study or provide informed consent (such as homelessness, drug/alcohol dependence, etc.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with a personal history of PCA; Unaffected males who are at higher risk for prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 595 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Family cancer history collection | Three years
  Collect detailed family cancer histories, personal medical history, prostate cancer clinical features, and exposure history from men with prostate cancer and men without prostate cancer to support studies focused on identifying hereditary cancer syndromes and genetic/epidemiologic factors predisposing to prostate cancer susceptibility.
Behavioral measure collection | Three years
  Collect behavioral measures to support research focused on assessing the needs of men undergoing cancer risk evaluation and satisfaction with the process
Biospecimen bank | Three years
  Create and maintain a biospecimen bank with specimens from men with prostate cancer and without prostate cancer to support studies focused on genetic alterations predisposing to prostate cancer risk
Genetic and genomic sequencing | Three years
  Perform targeted and broad-scale genetic and genomic sequencing to detect genetic alterations related to prostate cancer risk
Participant follow-up | Three years
  Develop mechanisms to recontact participants with updates on research genetic results to guide genetic testing for inherited prostate cancer risk.

CONTACTS AND LOCATIONS:
Overall Officials: Giri Veda, M.D., Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (3):
- United States (3):
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- See also: Sidney Kimmel Cancer Center — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/